CLINICAL TRIAL: NCT02033018
Title: Aflibercept Intravitreal Injection for Myopic Choroidal Neovascularization
Acronym: AflibxMyopia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JJ - 3/2013
Record Dates: First submitted 2013-12-31; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Choroidal Retinal Neovascularization
Keywords: Aflibercept; Myopia; Complications; Neovascularization; OCT
MeSH Terms: conditions — Myopia; Neovascularization, Pathologic | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept injection (Experimental): Myopic eyes with retinal neovascularization submitted a aflibercept intravitreal injection
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Aflibercept intravitreal injection
  Other Names: Aflibercept intravitreal injection of 0,5 mg ( 0.05mL

SUMMARY:
The purpose of this study is to evaluate the clinical results of anti-VEGF intra-vitreal injections (IVT) in CNV secondary

DETAILED DESCRIPTION:
Twenty consecutive patients (30 eyes) with subfoveal PM-CNV, 9 of whom had been unsuccessfully treated with Visudyne PDT, were treated with IVT of 0.5mg ranibizumab. ETDRS best corrected visual acuity, macular thickness on OCT scans, and angiographic features were recorded and evaluated. The aspect of OCT scans passing across the PM-CNV was also analyzed. IVTs were repeated only in case of persistent angiographic leakage and if OCT scans showed retinal thickening or edema and serous retinal detachment. The follow-up period was at least 6 months

ELIGIBILITY:
Inclusion Criteria:

* Myopic and CNVM

Exclusion Criteria:

* Patients with poor compliance
* Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications like recent history of Stroke or myocardial infraction (< one year). (Physician clearance was obtained for all patients).
* Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
* Patients who had undergone major surgery 28 days before, were excluded from the study and it was also suspended prior to elective surgery.
* Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
* Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR.
* Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy | To evaluate the clinical results of aflibercept intravitreal injection (AII) in choroidal neovascularization (CNV) secondary to pathologic myopia (PM-CNV), after 1 year follow up.
  8 patients with subfoveal PM-CNV, were treated with of 2 mg ( 0.05mL) RII. ETDRS best corrected visual acuity, macular thickness on OCT scans, and angiographic features were recorded and evaluated. The aspect of OCT scans passing across the PM-CNV was also analyzed. AII were repeated only in case of persistent angiographic leakage and if OCT scans showed retinal thickening or edema and serous retinal detachment. The follow-up period was at least 1 year.

SECONDARY OUTCOMES:
Safety and Tolerability | To evaluate the clinical results of aflibercept intravitreal injection (AII) in choroidal neovascularization (CNV) secondary to pathologic myopia (PM-CNV), after 1 year follow up.
  8 patients with subfoveal PM-CNV, were treated with of 2 mg ( 0.05mL) RII. ETDRS best corrected visual acuity, macular thickness on OCT scans, and angiographic features were recorded and evaluated. The aspect of OCT scans passing across the PM-CNV was also analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Joao J Nassaralla, Jr, Study Chair — Instituto de Olhos de Goiânia
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil